CLINICAL TRIAL: NCT01655732
Title: Effect of Atraumatic Restorative Treatment on Streptococcus Mutans Count in Saliva of Pregnant Women, A Randomized Control Trial
Brief Title: Effect of Atraumatic Restorative Treatment on Streptococcus Mutans Count in Saliva of Pregnant Women
Acronym: ART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheikh Zayed Federal Postgraduate Medical Institute (Other)
Collaborators: University of the Punjab (Other)
Responsible Party: Principal Investigator, Dr.Rabia Asad, Principal Investigator, Sheikh Zayed Federal Postgraduate Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rabia
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Pregnancy
Keywords: Pregnancy
MeSH Terms: interventions — Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atraumatic Restorative Treatment (Experimental): ART is Atraumatic Restorative Treatment involving removal of soft carious enamel and dentine by hand instruments only and then restore the resulting cavity and adjacent pits and fissures with an adhesive restorative material.
  Interventions: Procedure: Atraumatic Restorative Treatment

INTERVENTIONS:
Procedure: Atraumatic Restorative Treatment — ART is simple uninvasive technique involving removal of soft carious enamel and dentine by hand instrument only and then restore the cavity with adhesive restorative material.
  Other Names: ART

SUMMARY:
S. mutans counts have been found to be high in women with high level of untreated caries. In Pakistan 95% of all carious lesions are untreated that is an alarming situation. A majority of mother's have high level of caries and pose an increase risk of vertically transmitting it to their children. Therefore, the aim of this study is to determine the effect of A Traumatic Restorative Treatment(ART) in reducing S. mutans count in pregnant women and indirectly reduce the vertical transmission of S. mutans to their children so that ART as a preventive program may be provided and promoted in periurban areas where there is a lack of accessibility to oral health care.

DETAILED DESCRIPTION:
Dental caries is a multifactorial bacterial disease that is a significant public health problem in many countries.Microbiological and molecular studies show that there are increase chances of caries development in pregnant women.The reason is that Pregnancy is a condition involving many physical and physiological changes that may lead to many temporary adaptive changes in the body structure. This occurs due to release of number of hormones as estrogen, progesterone, relaxin and gonadotropin.

Studies using phenotyping and genotyping techniques have strongly proposed that mother is the primary source of infection for children who carry S. mutans strains and saliva is the main source of S. mutans transfer.The rate and degree of transmission depends on degree of infection of the parent, caretaker or playmate, the frequency of contact with the infant and his/her diet and immune status.Recent studies show that infants can get colonize by S. mutans from their mothers before the eruption of their primary teeth.

Hames et al (2006) has found that there is a positive correlation between the infected children and their parents with high S. mutans count.It was found that parents who had high levels of S. mutans in their saliva were the source of transmission of S. mutans in their children concluding that several preventive programs could be beneficial to prevent vertical transmission from mothers to infants.

Studies have also shown that preventive care measures in pregnant women or mother with younger children leads to reduction in S. mutans levels in them with subsequent decrease in colonization of these microorganisms and caries development.Recent research work has also reported that preventive program applied to the pregnant women reduce both the amount of plaque and S. mutans colonization and thus has a positive effect.

There are few interventional studies to determine the effect of oral environment stabilization (OES) procedure on S. mutans count in pregnant women through ART. Volpato et al (2011) found that there is a decrease in S. mutans colony forming units counts ,with a statistically significant difference (p<0.0001),between pregnant women's saliva samples before and after OES.And he concluded that OES is an effective clinical procedure in diminishing the number of Streptococcus mutans colony forming units in the saliva of high-caries risk pregnant women. This management is simple and effective, equivalent to the basic treatment needs of pregnant women that look for dental care in public service.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from enrolled population.
* Pregnant women having at least 3 untreated carious teeth.

Exclusion Criteria:

* Presence of any systemic diseases like diabetes, hypertension, cardiac disease.
* Deep carious lesions involving pulp.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Salivary s.mutans count | 6 months
  Atraumatic Restorative Treatment reduces the Streptococcus mutans count in oral flora of pregnant women that will indirectly reduces vertical transmission of Streptococcus mutans from mothers to infants.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Ayyaz A Khan, PhD, Study Director — Shaikh zayed Medical Complex
Locations (1):
- Shaikh Zayed Medical Complx, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Result] Volpato FC, Jeremias F, Spolidorio DM, Silva SR, Valsecki Junior A, Rosell FL. Effects of oral environment stabilization procedures on Streptococcus mutans counts in pregnant women. Braz Dent J. 2011;22(4):280-4. doi: 10.1590/s0103-64402011000400003. PMID 21861025